CLINICAL TRIAL: NCT06186336
Title: Feasibility of a Deep Learning-based Algorithm for Non-invasive Assessment of Vulnerable Coronary Plaque
Acronym: FOCUS DL
Status: Not yet recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Azienda Socio-Sanitaria Territoriale di Pavia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12019187648
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Chronic Coronary Syndrome; Coronary Artery Disease; Stable Angina; Acute Coronary Syndrome
Keywords: Coronary CT Angiography; Invasive Coronary Angiography; Optical Coherence Tomography; Vulnerable Coronary Plaque
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- DL-Based Vulnerable Plaque Detection and Assessment Tool: Enrolled subjects will receive a clinically indicated CCTA and ICA with OCT within 10 days. At least two qualified CCTA radiologists will independently review and annotate the coronary plaques in the CCTA using their local post-processing tools. At least two trained OCT readers will review and annotate the coronary plaques in the ICA/OCT using their local post-processing tools.
  The original de-identified CCTA data will be inputted into the Vulnerable Plaque Detection and Assessment Tool. The tool will perform the automatic identification of the plaque location and characteristics. These results will be compared to assess the algorithm's performance.
  Interventions: Other: Deep Learning-based Vulnerable Plaque Detection and Assessment Tool

INTERVENTIONS:
Other: Deep Learning-based Vulnerable Plaque Detection and Assessment Tool — Scanning requirements for the clinically indicated CCTA and ICA with OCT will be performed according to current site(s) guidelines and procedures. Administration of medications (such as contrast agents and potentially beta-blockers and other medications) will be given according to standard hospital care.
  This is a prospective research study evaluating an investigational product. The tool's use is intended for research purposes and is not intended as a substitute for required medical care. The CCTA and ICA with OCT will be processed in real-time using the site's locally available post-processing tools in order to guide the subject's medical care. Once the ICA with OCT is complete, the de-identified CCTA data will be inputted in the investigational tool.
  The clinically indicated CCTA and the ICA with OCT will both take approximately 1 hour and will take place within 10 days. No additional imaging is needed as part of the study.

SUMMARY:
The primary objective of this study is to assess the accuracy in terms of sensitivity, specificity, negative and positive predicted values of the DL-based algorithm with respect to correct identification of the plaque and associated vulnerability grade.

DETAILED DESCRIPTION:
Data collected in this study will be used for technology development, scientific evaluation, education, and regulatory submissions for future products. This is a pre-market, open label, prospective, non-randomized clinical research study conducted at one site in Italy. The product being researched is the Deep Learning-based (DL) algorithm for non-invasive detection of vulnerable coronary plaque.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for a clinically indicated CCTA and ICA with OCT imaging examinations;
2. Diagnosis of chronic coronary syndrome, known CAD, or stable angina; AND,
3. Patients with ACS that may undergo a CCTA and not refer directly to the Cath lab for revascularization procedures.

Exclusion Criteria:

1. Contradictions to contrast;
2. Contraindications for beta blocker;
3. BMI >30;
4. High heart rate ≥75 BPM;
5. Atrial Fibrillation;
6. Arrythmia or irregular heartbeats;
7. Any prior coronary revascularization;
8. Presence of pacemaker or implantable cardioverter defibrillator; OR,
9. Patients with TAVI/TAVR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with chronic coronary syndrome or stable angina, as well as patients with signs of acute coronary syndrome who have been ordered a clinically indicated CCTA and will likely be referred to undergo an ICA combined with OCT will be enrolled in this study. Subjects with recent onset or growing angina may be included in the study. Subjects will be representative of the general population expected to undergo cardiac non-invasive and invasive imaging and treatment procedures as standard of care clinical practice.
  The CCTA and ICA with OCT must be carried out within 10 days one from each other. Clinical decision for a PCI after the diagnostic procedures will not limit the enrollment. To preserve the aspect of the plaque, CCTA must be performed first.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Data Collection | Through study completion, an average of 1 year
  Number of subjects with raw CCTA and ICA with OCT data

SECONDARY OUTCOMES:
Accuracy of Tool | Through study completion, an average of 1 year
  Sensitivity, specificity, negative, and positive predicted values of the DL-based algorithm with respect to correct identification of the plaque and associated vulnerability grade in comparison to qualified readers
Safety Events | Through study completion, an average of 1 year
  Number of AEs, SAEs, and product issues

CONTACTS AND LOCATIONS:
Overall Officials: Paul Deak, Study Director — GE Healthcare
Locations (1):
- Ospedale Di Voghera, Azienda Socio-Sanitaria Territoriale di Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No